CLINICAL TRIAL: NCT04936282
Title: Treatment of Early Borderline Lesions in Low Immunological Risk Kidney Transplant Patients: a Spanish Multicenter, Randomized, Controlled Parallel-group Trial: The TRAINING Study
Brief Title: Treatment of Early Borderline Lesions in Low Immunological Risk Kidney Transplant Patients (TRAINING)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Canaria de Investigación Sanitaria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRAINING
Record Dates: First submitted 2021-06-18; First posted 2021-06-23 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Kidney Transplant Failure and Rejection
Keywords: borderline lesions; α-klotho; low immunological risk; subclinical inflammation; kidney transplant
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Normal treatment (Steroids, tacrolimus and mycophenolate) for first 90 days, then add Grafalon single-dose if borderline lesions are present in protocol biopsy (performed at third month post-transplantation).
  Interventions: Drug: Grafalon
- Normal treatment (Active Comparator): Normal treatment (Steroids, tacrolimus and mycophenolate) arm
  Interventions: Drug: Normal Treatment

INTERVENTIONS:
Drug: Grafalon — When Borderline lesions are present in protocol biopsy, administer Grafalon ® 6 mg/kg/day in a single day. Then continue with the normal treatment: Steroids (5 mg/day), tacrolimus (0.1 mg/kg/day) and mycophenolate (1000 mg/day).
  Arms: Experimental
Drug: Normal Treatment — When Borderline lesions are present in protocol biopsy, administer the normal treatment: Steroids (5 mg/day), tacrolimus (0.1 mg/kg/day) and mycophenolate (1000 mg/day)
  Arms: Normal treatment

SUMMARY:
Background: Subclinical inflammation, including borderline lesions (BL), is very common (30-40%) after kidney transplantation (KT), even in low immunological risk patients, and can lead to interstitial fibrosis/tubular atrophy (IFTA) and worsening of renal function with graft loss. Few controlled studies have analyzed the therapeutic benefit of these BL on renal function and graft histology. Furthermore, these studies have only used bolus steroids, which may be insufficient to slow the progression of these lesions. Klotho, a transmembrane protein produced mainly in the kidney with antifibrotic properties, plays a crucial role in the senescence-inflammation binomial of kidney tissue. Systemic and local inflammation decrease renal tissue expression and soluble levels of α-klotho. It is therefore important to determine whether treatment of BL prevents a decrease in α klotho levels, progression of IFTA, and loss of kidney function.

Methods: The TRAINING study will randomize 80 patients with low immunological risk who will receive their first KT. The aim of the study is to determine whether the treatment of early BL (3rd month post-KT) with polyclonal rabbit antithymocyte globulin (Grafalon®) (6 mg/kg/day) prevents or decreases the progression of IFTA and the worsening of graft function compared to conventional therapy after two years post-TX, as well as to analyze whether treatment of BL with Grafalon® can modify the expression and levels of klotho, as well as the pro-inflammatory cytokines that regulate its expression.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex, older than 18 years, with no immunological risk (PRA<20% and absence of DSA), who receive their first deceased donor or living donor KT.
* Presence of BL, excluding isolated inflammation (t0, i>0) and isolated tubulitis (t>0, i0).
* Patients receiving tacrolimus in combination with mycophenolic acid (MPA) and steroids.
* Absence of clinical or subclinical and histological immunological dysfunction before randomization.
* Absence of de novo DSA anti-HLA antibodies at the time of randomization.
* Provision of written informed consent.
* Acceptance of efficient contraception in women.

Exclusion Criteria:

* Recipients of a multi-organ transplant.
* Re-transplants.
* Patients without inflammation in the third month protocol biopsy (i0,t0), or with isolated inflammation without tubulitis (t0,i>0) or isolated tubulitis without inflammation (t>0,i0).
* Presence of DSA antibodies before transplantation or at randomization.
* Cold ischemia time >30 hours.
* Serum creatinine >2.5 mg/dl or proteinuria >1 g/day at randomization.
* Presence of significant thrombopenia (<100,000/mm3) or leukopenia (<3000 mm/3) at randomization.
* Previous episode of clinical or subclinical rejection (≥IA) before randomization.
* CMV disease in the first three months after transplantation.
* BK-polyomavirus nephropathy at randomization.
* Recurrent or de novo glomerulonephritis.
* Treatment with immunosuppressive drugs other than those in this clinical trial.
* Patients who are positive for the human immunodeficiency virus (HIV) or with severe systemic infection, who, in the opinion of the investigator, require continued therapy.
* Previous (within the last 5 years) or present malignancy, except excised basal or squamous cell carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Presence of interstitial fibrosis/tubular atrophy (IFTA) | 24 months
  Measurement at 24 months according to the Banff classification. The Banff Classification of Allograft Pathology is an international consensus classification for the reporting of biopsies from solid organ transplant.
Renal function measured with CKD-EPI | 24 months
  Renal function after kidney transplant in both groups at 24 months measured according to glomerular filtration rate determined by CKD-EPI formula

SECONDARY OUTCOMES:
Graft Survival | 24 months
  Graft survival after kidney transplant in both groups
Patient Survival | 24 months
  Patient survival after kidney transplant in both groups
Assess the Adherence to Immunosuppressive Therapy in the Two Treatment Groups | 24 months
  The Basle scale was used to assess adherence to immunosuppressive therapy.
Incidence of Diabetes Mellitus | 24 months
  Incidence of diabetes mellitus after kidney transplant in both groups at 1, 2, 3, 4, 6, 9, 12, 18 and 24 months
Blood Pressure mmHg | 24 months
  Blood pressure after kidney transplant in both groups at 24 months
Number of Participants With Acute Rejection Lesions | 24 months
  Patients with acute rejection lesions (including subclinical rejection) at 24 months according to Banff classification
Lipid Profile cholesterol, triglycerides | 24 months
  Lipid profile after kidney transplant in both groups at 24 months
Klotho levels pg/ml | 24 months
  Klotho levels after kidney transplant in both groups at 1, 3, 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, None Selected
  - Fundación Puigvert, Barcelona
  - Hospital Universitari Valld´Hebron, Barcelona
  - Veronica Lopez Jimenez, Málaga

REFERENCES:
- [Background] Riella LV, Djamali A, Pascual J. Chronic allograft injury: Mechanisms and potential treatment targets. Transplant Rev (Orlando). 2017 Jan;31(1):1-9. doi: 10.1016/j.trre.2016.10.005. Epub 2016 Oct 11. PMID 27847221
- [Background] Kasiske BL, Gaston RS, Gourishankar S, Halloran PF, Matas AJ, Jeffery J, Rush D. Long-term deterioration of kidney allograft function. Am J Transplant. 2005 Jun;5(6):1405-14. doi: 10.1111/j.1600-6143.2005.00853.x. PMID 15888048
- [Background] Nankivell BJ, Borrows RJ, Fung CL, O'Connell PJ, Allen RD, Chapman JR. The natural history of chronic allograft nephropathy. N Engl J Med. 2003 Dec 11;349(24):2326-33. doi: 10.1056/NEJMoa020009. PMID 14668458
- [Background] Garcia-Carro C, Dorje C, Asberg A, Midtvedt K, Scott H, Reinholt FP, Holdaas H, Seron D, Reisaeter AV. Inflammation in Early Kidney Allograft Surveillance Biopsies With and Without Associated Tubulointerstitial Chronic Damage as a Predictor of Fibrosis Progression and Development of De Novo Donor Specific Antibodies. Transplantation. 2017 Jun;101(6):1410-1415. doi: 10.1097/TP.0000000000001216. PMID 27163535
- [Background] Ortiz F, Gelpi R, Helantera I, Melilli E, Honkanen E, Bestard O, Grinyo JM, Cruzado JM. Decreased Kidney Graft Survival in Low Immunological Risk Patients Showing Inflammation in Normal Protocol Biopsies. PLoS One. 2016 Aug 17;11(8):e0159717. doi: 10.1371/journal.pone.0159717. eCollection 2016. PMID 27532630
- [Background] Rush DN, Gibson IW. Subclinical Inflammation in Renal Transplantation. Transplantation. 2019 Jun;103(6):e139-e145. doi: 10.1097/TP.0000000000002682. PMID 30801537
- [Background] Nankivell BJ, Agrawal N, Sharma A, Taverniti A, P'Ng CH, Shingde M, Wong G, Chapman JR. The clinical and pathological significance of borderline T cell-mediated rejection. Am J Transplant. 2019 May;19(5):1452-1463. doi: 10.1111/ajt.15197. Epub 2019 Jan 22. PMID 30501008
- [Background] Moreso F, Ibernon M, Goma M, Carrera M, Fulladosa X, Hueso M, Gil-Vernet S, Cruzado JM, Torras J, Grinyo JM, Seron D. Subclinical rejection associated with chronic allograft nephropathy in protocol biopsies as a risk factor for late graft loss. Am J Transplant. 2006 Apr;6(4):747-52. doi: 10.1111/j.1600-6143.2005.01230.x. PMID 16539631
- [Background] Mehta RB, Tandukar S, Jorgensen D, Randhawa P, Sood P, Puttarajappa C, Zeevi A, Tevar AD, Hariharan S. Early subclinical tubulitis and interstitial inflammation in kidney transplantation have adverse clinical implications. Kidney Int. 2020 Aug;98(2):436-447. doi: 10.1016/j.kint.2020.03.028. Epub 2020 Apr 25. PMID 32624181
- [Background] Mehta R, Bhusal S, Randhawa P, Sood P, Cherukuri A, Wu C, Puttarajappa C, Hoffman W, Shah N, Mangiola M, Zeevi A, Tevar AD, Hariharan S. Short-term adverse effects of early subclinical allograft inflammation in kidney transplant recipients with a rapid steroid withdrawal protocol. Am J Transplant. 2018 Jul;18(7):1710-1717. doi: 10.1111/ajt.14627. Epub 2018 Jan 17. PMID 29247472
- [Background] Loupy A, Haas M, Roufosse C, Naesens M, Adam B, Afrouzian M, Akalin E, Alachkar N, Bagnasco S, Becker JU, Cornell LD, Clahsen-van Groningen MC, Demetris AJ, Dragun D, Duong van Huyen JP, Farris AB, Fogo AB, Gibson IW, Glotz D, Gueguen J, Kikic Z, Kozakowski N, Kraus E, Lefaucheur C, Liapis H, Mannon RB, Montgomery RA, Nankivell BJ, Nickeleit V, Nickerson P, Rabant M, Racusen L, Randhawa P, Robin B, Rosales IA, Sapir-Pichhadze R, Schinstock CA, Seron D, Singh HK, Smith RN, Stegall MD, Zeevi A, Solez K, Colvin RB, Mengel M. The Banff 2019 Kidney Meeting Report (I): Updates on and clarification of criteria for T cell- and antibody-mediated rejection. Am J Transplant. 2020 Sep;20(9):2318-2331. doi: 10.1111/ajt.15898. Epub 2020 May 28. PMID 32463180
- [Background] Beimler J, Zeier M. Borderline rejection after renal transplantation--to treat or not to treat. Clin Transplant. 2009 Dec;23 Suppl 21:19-25. doi: 10.1111/j.1399-0012.2009.01105.x. PMID 19930312
- [Background] Kee TY, Chapman JR, O'Connell PJ, Fung CL, Allen RD, Kable K, Vitalone MJ, Nankivell BJ. Treatment of subclinical rejection diagnosed by protocol biopsy of kidney transplants. Transplantation. 2006 Jul 15;82(1):36-42. doi: 10.1097/01.tp.0000225783.86950.c2. PMID 16861939
- [Background] Park SH, Friedewald JJ. Are borderline changes real rejection? Current viewpoints. Curr Opin Nephrol Hypertens. 2020 Nov;29(6):656-662. doi: 10.1097/MNH.0000000000000648. PMID 32889982
- [Background] Opelz G, Naujokat C, Daniel V, Terness P, Dohler B. Disassociation between risk of graft loss and risk of non-Hodgkin lymphoma with induction agents in renal transplant recipients. Transplantation. 2006 May 15;81(9):1227-33. doi: 10.1097/01.tp.0000219817.18049.36. PMID 16699447
- [Background] Brennan DC, Daller JA, Lake KD, Cibrik D, Del Castillo D; Thymoglobulin Induction Study Group. Rabbit antithymocyte globulin versus basiliximab in renal transplantation. N Engl J Med. 2006 Nov 9;355(19):1967-77. doi: 10.1056/NEJMoa060068. PMID 17093248
- [Background] Oostenbrink LVE, Jol-van der Zijde CM, Kielsen K, Jansen-Hoogendijk AM, Ifversen M, Muller KG, Lankester AC, van Halteren AGS, Bredius RGM, Schilham MW, van Tol MJD. Differential Elimination of Anti-Thymocyte Globulin of Fresenius and Genzyme Impacts T-Cell Reconstitution After Hematopoietic Stem Cell Transplantation. Front Immunol. 2019 Mar 6;10:315. doi: 10.3389/fimmu.2019.00315. eCollection 2019. PMID 30894854
- [Background] Shimony O, Nagler A, Gellman YN, Refaeli E, Rosenblum N, Eshkar-Sebban L, Yerushalmi R, Shimoni A, Lytton SD, Stanevsky A, Or R, Naor D. Anti-T lymphocyte globulin (ATG) induces generation of regulatory T cells, at least part of them express activated CD44. J Clin Immunol. 2012 Feb;32(1):173-88. doi: 10.1007/s10875-011-9599-2. Epub 2011 Oct 7. PMID 21979414
- [Background] Izquierdo MC, Perez-Gomez MV, Sanchez-Nino MD, Sanz AB, Ruiz-Andres O, Poveda J, Moreno JA, Egido J, Ortiz A. Klotho, phosphate and inflammation/ageing in chronic kidney disease. Nephrol Dial Transplant. 2012 Dec;27 Suppl 4:iv6-10. doi: 10.1093/ndt/gfs426. PMID 23258814
- [Background] Kim HR, Nam BY, Kim DW, Kang MW, Han JH, Lee MJ, Shin DH, Doh FM, Koo HM, Ko KI, Kim CH, Oh HJ, Yoo TH, Kang SW, Han DS, Han SH. Circulating alpha-klotho levels in CKD and relationship to progression. Am J Kidney Dis. 2013 Jun;61(6):899-909. doi: 10.1053/j.ajkd.2013.01.024. Epub 2013 Mar 27. PMID 23540260
- [Background] Zhou L, Mo H, Miao J, Zhou D, Tan RJ, Hou FF, Liu Y. Klotho Ameliorates Kidney Injury and Fibrosis and Normalizes Blood Pressure by Targeting the Renin-Angiotensin System. Am J Pathol. 2015 Dec;185(12):3211-23. doi: 10.1016/j.ajpath.2015.08.004. Epub 2015 Oct 24. PMID 26475416
- [Background] Otani-Takei N, Masuda T, Akimoto T, Honma S, Watanabe Y, Shiizaki K, Miki T, Kusano E, Asano Y, Kuro-O M, Nagata D. Association between Serum Soluble Klotho Levels and Mortality in Chronic Hemodialysis Patients. Int J Endocrinol. 2015;2015:406269. doi: 10.1155/2015/406269. Epub 2015 Oct 28. PMID 26604925
- [Background] Ruiz-Andres O, Sanchez-Nino MD, Moreno JA, Ruiz-Ortega M, Ramos AM, Sanz AB, Ortiz A. Downregulation of kidney protective factors by inflammation: role of transcription factors and epigenetic mechanisms. Am J Physiol Renal Physiol. 2016 Dec 1;311(6):F1329-F1340. doi: 10.1152/ajprenal.00487.2016. Epub 2016 Oct 19. PMID 27760772
- [Background] Moreno JA, Izquierdo MC, Sanchez-Nino MD, Suarez-Alvarez B, Lopez-Larrea C, Jakubowski A, Blanco J, Ramirez R, Selgas R, Ruiz-Ortega M, Egido J, Ortiz A, Sanz AB. The inflammatory cytokines TWEAK and TNFalpha reduce renal klotho expression through NFkappaB. J Am Soc Nephrol. 2011 Jul;22(7):1315-25. doi: 10.1681/ASN.2010101073. Epub 2011 Jun 30. PMID 21719790
- [Background] Nankivell BJ, P'Ng CH, Chapman JR. Does tubulitis without interstitial inflammation represent borderline acute T cell mediated rejection? Am J Transplant. 2019 Jan;19(1):132-144. doi: 10.1111/ajt.14888. Epub 2018 Jun 15. PMID 29687946
- [Background] Srinivas TR, Meier-Kriesche HU. Minimizing immunosuppression, an alternative approach to reducing side effects: objectives and interim result. Clin J Am Soc Nephrol. 2008 Mar;3 Suppl 2(Suppl 2):S101-16. doi: 10.2215/CJN.03510807. PMID 18308998
- [Background] Xu C, Chang A, Hack BK, Eadon MT, Alper SL, Cunningham PN. TNF-mediated damage to glomerular endothelium is an important determinant of acute kidney injury in sepsis. Kidney Int. 2014 Jan;85(1):72-81. doi: 10.1038/ki.2013.286. Epub 2013 Jul 31. PMID 23903370
- [Background] Sharif MN, Campanholle G, Nagiec EE, Wang J, Syed J, O'Neil SP, Zhan Y, Brenneman K, Homer B, Neubert H, Karim R, Pullen N, Evans SM, Fleming M, Chockalingam P, Lin LL. Soluble Fn14 Is Detected and Elevated in Mouse and Human Kidney Disease. PLoS One. 2016 May 12;11(5):e0155368. doi: 10.1371/journal.pone.0155368. eCollection 2016. PMID 27171494
- [Background] Park WD, Griffin MD, Cornell LD, Cosio FG, Stegall MD. Fibrosis with inflammation at one year predicts transplant functional decline. J Am Soc Nephrol. 2010 Nov;21(11):1987-97. doi: 10.1681/ASN.2010010049. Epub 2010 Sep 2. PMID 20813870
- [Background] Kurtkoti J, Sakhuja V, Sud K, Minz M, Nada R, Kohli HS, Gupta KL, Joshi K, Jha V. The utility of 1- and 3-month protocol biopsies on renal allograft function: a randomized controlled study. Am J Transplant. 2008 Feb;8(2):317-23. doi: 10.1111/j.1600-6143.2007.02049.x. Epub 2007 Dec 18. PMID 18093273
- [Derived] Hernandez D, Vazquez-Sanchez T, Sola E, Lopez V, Ruiz-Esteban P, Caballero A, Salido E, Leon M, Rodriguez A, Serra N, Rodriguez C, Facundo C, Perello M, Silva I, Marrero-Miranda D, Cidraque I, Moreso F, Guirado L, Seron D, Torres A. Treatment of early borderline lesions in low immunological risk kidney transplant patients: a Spanish multicenter, randomized, controlled parallel-group study protocol: the TRAINING study. BMC Nephrol. 2022 Nov 7;23(1):357. doi: 10.1186/s12882-022-02989-z. PMID 36344929